CLINICAL TRIAL: NCT06894797
Title: The Efficacy and Safety of Long-Course Preoperative Chemoradiotherapy Combined With Consolidation or Induction NALIRIFOX Chemotherapy in the Treatment of Locally Advanced Rectal Cancer: A Prospective, Multicenter, Phase II Study.
Brief Title: Preoperative Chemoradiotherapy Combined With Consolidation or Induction NALIRIFOX in Rectal Cancer.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yongheng Li, Director, Peking University Cancer Hospital & Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DNY- LARC-BJ01
Record Dates: First submitted 2025-03-12; First posted 2025-03-25 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Rectal Cancer
MeSH Terms: interventions — Capecitabine; irinotecan sucrosofate; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long-Course Preoperative Chemoradiotherapy Combined with Consolidation NALIRIFOX Chemotherapy (Experimental): Patients will receive Concurrent Chemoradiotherapy（Radiation + Capecitabine） followed by NALIRIFOX
  Concurrent Chemoradiotherapy：5 Weeks in total
  NALIRIFOX：8 Weeks in total
  Interventions: Radiation: Concurrent Chemoradiotherapy（Radiation + Capecitabine）; Drug: irinotecan hydrochloride liposome injection; Drug: Oxaliplatin; Drug: 5-FU
- Long-Course Preoperative Chemoradiotherapy Combined with Induction NALIRIFOX Chemotherapy (Experimental): Patients will receive NALIRIFOX followed by Concurrent Chemoradiotherapy（Radiation + Capecitabine）
  Concurrent Chemoradiotherapy：5 Weeks in total
  NALIRIFOX：8 Weeks in total
  Interventions: Radiation: Concurrent Chemoradiotherapy（Radiation + Capecitabine）; Drug: irinotecan hydrochloride liposome injection; Drug: Oxaliplatin; Drug: 5-FU

INTERVENTIONS:
Radiation: Concurrent Chemoradiotherapy（Radiation + Capecitabine） — Capecitabine 825 mg/m^2 Po BlD, Monday-Friday, on days of radiation treatment only, throughout the duration of RT Radiation：45-50Gy/25fractions/5 weeks，5fractions/week
Drug: irinotecan hydrochloride liposome injection — Irinotecan hydrochloride liposome injection (50mg/m^2) will be administered by intravenous infusion on day 1 in a 2-week treatment cycle.
  Other Names: Nal-IRI
Drug: Oxaliplatin — Oxaliplatin (60mg/m^2) will be administered by intravenous infusion on day 1 in a 2-week treatment cycle.
  Other Names: OXA
Drug: 5-FU — 5-FU (2400mg/m^2) will be administered by intravenous infusion on 46h in a 2-week treatment cycle.
  Other Names: fluorouracil

SUMMARY:
The Efficacy and Safety of Long-Course Preoperative Chemoradiotherapy Combined with Consolidation or Induction NALIRIFOX Chemotherapy in the Treatment of Locally Advanced Rectal Cancer: A Prospective, Multicenter, Phase II Study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects participate in the study need to sign the informed consent, and demonstrate good compliance.
2. Age: 18~75 years old.
3. Histopathologically confirmed rectal adenocarcinoma.
4. Locally advanced rectal cancer, determined at baseline.
5. No prior systemic therapy.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0~1.
7. Expected survival ≥ 12 months.
8. Adequate bone marrow function (In the absence of blood transfusion within 14 days, correction with granulocyte colony-stimulating factor or other hematopoietic stimulating factor was not used within 7 days prior to laboratory examination) :

   ①Absolute neutrophil count (ANC) ≥1.5×10^9/L, Platelet count ≥100×10^9/L, Hemoglobin (Hb) ≥9g/dL.

   ② Liver function: Total bilirubin ≤1.5 × upper limit of normal (ULN), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN, liver metastasis, AST and ALT≤5×ULN.

   ③ Renal function: Serum creatinine (Cr) ≤1.5 × ULN or creatinine clearance ≥60 mL/min.

   ④International Normalized Ratio (INR) ≤ 1.5 ULN, Prothrombin time and activated partial thromboplastin time (APTT) ≤ 1.5 ULN
9. Microsatellite Stability (MSS) or proficient MisMatch Repair (pMMR).

Exclusion Criteria:

1. Within 4 weeks prior to treatment, subjects must not have received radiotherapy, surgery, chemotherapy, immunotherapy for tumors, molecular targeted therapies, or other investigational drugs.
2. microsatellite instability (MSI) or mismatch repair gene deletion (dMMR)
3. Distant metastasis
4. Significant clinical bleeding symptoms or significant bleeding tendency within 3 months prior to treatment (bleeding > 30ml within 3 months), hematemesis, black stool, blood in the stool), hemoptysis (> 5 mL of fresh blood within 4 weeks), etc. Treatment of venous/venous thrombotic events within the first 6 months, such as cerebrovascular accidents (including transient brain lesions) Ischemic attack, cerebral hemorrhage, cerebral infarction), deep vein thrombosis and pulmonary embolism; Or need to use warfarin or Long-term anticoagulant therapy with heparin, or long-term antiplatelet therapy (aspirin ≥300 mg/day or chlorine) is required Picogrel ≥75 mg/day).
5. During screening, tumors were found to invade large vascular structures, such as pulmonary artery, superior vena cava or inferior vena cava that there was a risk of major bleeding by the investigator judged.
6. Active heart disease, including myocardial infarction, severe/unstable angina, occurred 6 months before treatment. ultrasonic Left ventricular ejection fraction <50% was detected by cardiogram, indicating poor arrhythmia control.
7. High blood pressure that is not well controlled by antihypertensive medication (systolic blood pressure ≥140 mmHg and/or diastolic pressure ≥90 mmHg).
8. Any other malignancy within 5 years, with the exception of cured in-situ carcinoma or basal cell carcinoma etc.
9. Known or suspected allergy to the investigational drug or a similar drug.
10. Active or uncontrolled severe infection.
11. Known human immunodeficiency virus (HIV) infection.
12. Any other disease with clinically significant metabolic abnormalities, physical abnormalities, or laboratory abnormalities Often, in the investigator's judgment, there is reason to suspect that the patient has a disease or condition that is not suitable for use of the investigational drug state (such as having a seizure and requiring treatment) that will either affect the interpretation of the study results or make the patient In a high-risk situation.
13. Patients who have been co-administered a potent CYP3A4 inducer within 3 weeks prior to first dosing, or a potent CYP3A4 inhibitor or a potent UGT1A1 inhibitor within 3 weeks prior to first dosing
14. Inability to comply with study protocols or study procedures.
15. Patients who are not suitable to participate in this trial judged by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate | From baseline up to approximately 3 months
  To evaluate the efficacy of anti-tumor

CONTACTS AND LOCATIONS:
Overall Officials: Yongheng Li, MD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, China